CLINICAL TRIAL: NCT01841073
Title: Effect of Fermentable Carbohydrate on Glucose Homeostasis and Weight Management in Subjects With Prediabetes
Brief Title: Effect of Fermentable Carbohydrate on Glucose Homeostasis
Acronym: FermCarb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FermCarb
Record Dates: First submitted 2013-04-05; First posted 2013-04-26 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Prediabetes
Keywords: Prediabetes; Fermentable carbohydrate; Appetite; Glucose homeostasis; Weight management
MeSH Terms: conditions — Prediabetic State | interventions — Inulin; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin (Experimental): Subject will take 10g inulin for 2 weeks, 20g of inulin for the next 2 weeks and then 30g for the remainder of the investigations.
  Interventions: Dietary Supplement: Inulin
- Cellulose (Placebo Comparator): Subjects will take 10g cellulose a day for 2 weeks, followed by 20g a day for 2 weeks, then 30g a day for the rest of the study.
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Dietary Supplement: Inulin — Subjects will have 4 dietary counselling sessions in the first 9 weeks of the study with a goal to lose 5% of their body weight by week 9. They will be asked to maintain their weight loss until week 18.
  Other Names: Synergy1
  Arms: Inulin
Dietary Supplement: Cellulose — Subjects will have 4 dietary counselling sessions in the first 9 weeks of the study with a goal to lose 5% of their body weight by week 9. They will be asked to maintain their weight loss until week 18.
  Arms: Cellulose
Dietary Supplement: Inulin — Subject will take inulin for 6 weeks in total with no other change to their diet or lifestyle.
  Other Names: Synergy1
  Arms: Inulin
Dietary Supplement: Cellulose — Subject will take cellulose for 6 weeks in total with no other change to their diet or lifestyle.
  Arms: Cellulose
Dietary Supplement: Inulin — Subject will take inulin for 6 weeks in total with no other change to their diet or lifestyle.
  Subject will wear a Continuous Glucose Monitor for 4 x 5 days during the study.
  Other Names: Synergy1
  Arms: Inulin
Dietary Supplement: Cellulose — Subject will take cellulose for 6 weeks in total with no other change to their diet or lifestyle.
  Subject will wear a Continuous Glucose Monitor for 4 x 5 days during the study.
  Arms: Cellulose

SUMMARY:
The rise in the prevalence of type 2 diabetes is related to recent lifestyle changes leading to a rise in obesity. Obesity is a risk factor for Impaired Glucose Tolerance (IGT) and diabetes. A type of fibre - fermentable carbohydrate - may help prevent diabetes in individuals with IGT by reducing appetite and food intake, and improving insulin sensitivity. Although fermentable carbohydrate is not absorbed in the small intestine it is full fermented by the colonic bacteria. The fermentation of this carbohydrate produces short chain fatty acids which act on specific G protein coupled receptors (GPR41/43) in the intestine to release GLP-1 and PYY. GLP-1 and PYY are hormones which act on appetite centres in the brain to decrease appetite. GLP-1 incretin effects and possible effect of the beta cell will increase insulin sensitivity. Short chain fatty acids also suppress the release of free fatty acids from adipocytes. Lower levels of free fatty acids in insulin resistant subject's leads to improved insulin sensitivity. This body of work will examine the effect of fermentable carbohydrate on appetite, weight loss, blood glucose control which will give an indication of the possibility of fermentable carbohydrate to prevent type 2 diabetes in this at-risk group.

DETAILED DESCRIPTION:
TITLE The Effect of Fermentable Carbohydrate on Weight Management and Glycaemic Control in People at High Risk of Developing DMT2

AIMS To assess the effect of fermentable carbohydrate in subjects with pre-diabetes on:

1. Appetite regulation
2. Glucose homeostasis and B-cell function
3. Weight loss and changes in body composition
4. Weight loss maintenance
5. Markers of Oxidative Stress

DESIGN The investigators plan to conduct 3 investigations. Investigation 1 and 2 are Randomised Crossover Control Trials of 14 days supplementation with 30g of inulin (fermentable carbohydrate) or a cellulose (non fermentable carbohydrate) control to firstly describe the physiology and mechanisms behind appetite regulation and glucose homeostasis. Investigation 3 is a Randomised Control Parallel Study of weight loss followed by weight maintenance to assess the efficacy of fermentable carbohydrate to decrease risk of T2DM.

POPULATION Overweight and obese men or women with pre-diabetes.

TREATMENT Participants in the treatment arm in all 3 investigations will consume inulin 3 times per day (total daily dose: 30g). Participants in the placebo arm in all 3 investigations will be taking cellulose 3 times a day (total daily dose: 30g).

DURATION Investigation 1 will last 16 weeks. Investigation 2 will last 18 weeks. Investigation 3 will last 18 weeks.

BACKGROUND

Type 2 Diabetes (DMT2) is a major health concern in the UK, as it is worldwide. The increased prevalence of DMT2 in the UK is closely linked with the increased prevalence of obesity, with the risk for diabetes estimated to increase by 4.5-9 percent with every kilogram weight gained (1). Pre-diabetes is also associated with an increase in body weight, and is a critical step in the development of T2DM.

Having pre-diabetes also increases the risk for cardiovascular disease. It is thought this is due to the hyperglycaemia and glycaemic variability seen in the pre-diabetic state. Both hyperglycaemia and glycaemic variability are associated with oxidative stress. Oxidative stress is postulated to cause endothelial damage which can lead to cardiovascular disease. Reductions in hyperglycaemia and glycaemic variability may cause a reduction in oxidative stress.

A number of gut hormones - released physiologically in response to food - have been shown to powerfully inhibit human appetite and inhibit food intake and glucose homeostasis (2). Two of these gut hormones, glucagon like peptide-1 (GLP-1) and peptide YY (PYY) are released from the neuroendocrine L-cell in the colon, and have demonstrable appetite suppressive effects in animals and humans (3-6). GLP-1 also improves glycaemic control by stimulating pancreatic B-cells to secrete insulin in a glucose-dependent manner, inhibits glucagon release and reduces hepatic glucose output (7-9). Long-term treatment with GLP-1 agonists has been shown to cause significant weight loss in humans (10).

Work by ourselves and others in rodents have shown that dietary fermentable carbohydrates (FCHOs) can significantly increase circulating PYY and GLP-1 levels while suppressing appetite centres in the hypothalamus (11-12). This results in lower body fat and abdominal fat with no overall effect on weight; however as abdominal fat is an important cardiovascular risk factor in diabetes, this effect is likely to be favourable to health (13-14). In humans, there are a number of short-term studies that report an increase in satiety following consumption of FCHOs (15-16)and a year-long study of children consuming the FCHO inulin showed significant weight loss compared to controls (17). FCHO has also been shown to increase insulin sensitivity, reduce post-prandial blood glucose levels and enhance lipid oxidation in overweight subjects with and without diabetes (18,19), effects that may be mediated by the FCHO induced GLP-1 increase (GLP-1 was not measured in these studies). Even short-term consumption of FCHO in healthy subjects has a similar effect on glycaemic control (20).

STUDY DESIGN

Inulin will be used as the FCHO supplement in all 3 investigations. Inulin has no known effect on the small bowel, being fully fermented in the large bowel. Inulin is therefore ideally suited for the investigation of large bowel fermentation on human appetite, glycaemic control and weight maintenance. Test

SCREENING PROCEDURE

1. Telephone screening will identify the members of this cohort who meet the initial screening criteria of:

   Adults over 18 years of age, Participants with no major metabolic disease - including diabetes, no known/diagnosed gastrointestinal problem such as inflammatory bowel disease, irritable bowel syndrome etc and no drug or alcohol abuse in the last 2 years.
2. At the Sir John McMichael Centre, participants will undergo the following:

An oral glucose tolerance test.

A blood sample of 30ml will be taken for full blood count, liver function tests, electrolytes, thyroid function tests, HbA1c, and glucose.

Body weight and height will be recorded.

DETAILED PROTOCOL

APPETITE STUDY SESSIONS

Visit 1, 2, 3 & 4 in Investigation 1.

Participants arrive fasted overnight (10 hour fast). After explanation of the procedures and confirmation that the participant is happy to proceed, body weight is recorded.

A cannula is inserted in a forearm vein facilitating blood sampling throughout the day. Two baseline blood samples are withdrawn. Visual analogue scales (VAS) are completed every time a blood sample is drawn. The sampling scheme is presented below. A total of 80ml of blood will taken during investigation 1 appetite study days, and a total of 115ml be withdrawn during each appetite study visit in investigation 3. Visual Analogue scales to assess appetite will be completed each time a blood sample is taken. The Visual Analogue Scale questions include: "How full do you feel right now?" and "How hungry do you feel right now?" and "How much could you eat right now?". They will answer by making a vertical mark on a ten centimetre line anchored with the terms "not at all" and "extremely". Similarly, side-effects such as nausea, sickness, flatulence, bloating, diarrhoea, and general well-being will be assessed.

At time 0, breakfast is served and participants will have 20 minutes to consume the meal. Lunch is served at 240 minutes, and the meal test is served at 440 minutes after the last blood sample is taken.

During the study session, participants will be asked to minimize physical activity. Water is allowed freely, though participants will be requested not to drink less than 10 minutes prior to a blood sample and VAS completion. At 440 minutes, a pre-weighed meal is served. The meal is served in excess and participants are asked to eat until comfortably full. A jug of water is served with the meal and the water intake will also be recorded.

In investigation 3, the study sessions will be shorter, consisting of a breakfast and a meal test at lunch.

ONE TO ONE DIETARY COUNSELLING

In Investigation 3, all participants will receive dietary counselling at weeks 1, 2, 4, and 7. The instruction given to the participants will be individualised based on current weight and energy requirements, consistent with the usual package of care that would be offered within a dietitian clinic. The participants will be instructed to aim for 5% weight loss over 9 weeks.

SUPPLEMENTATION UNDER FREE-LIVING CONDITIONS

The supplement will be provided in sachets (containing 10g portions). During the run-in period the daily intake will gradually be increased to 30g per day over 4 weeks. During this run-in period the investigators will contact the participants via e-mail or telephone twice to ensure the fibre supplementation has no un-toward side-effects and ensure that instructions are followed and answer any questions the participants may have. The subjects then take 30g a day until the end of the study (at 6 weeks for investigation 1 or 18 weeks in investigation 3).

WASHOUT PERIOD

In investigations 1 and 2 there will be a wash out period of 4 weeks before the subject crosses over the the alternate supplementation.

DIETARY RECORDS, APPETITE AND SIDE-EFFECTS

A 3-day dietary record is to be completed for the 3 days preceding visits 1, 2 and 3 during Investigation 1, and visits 1, 6 and 7 during Investigation 3. On the same days, appetite sensation and side-effects will be assessed using visual analogue scales. The Visual Analogue Scale questions include: "How full did you feel after eating meals today?" and "How hungry did you feel between meals today?". They will answer by making a vertical mark on a ten centimetre line anchored with the terms "not at all" and "extremely". Similarly, side-effects such as nausea, sickness, flatulence, bloating, diarrhoea, and general well-being will be assessed.

METHODS FOR ASSESSING INSULIN AND GLUCOSE HOMOSTASIS MEAL TOLERANCE TEST Participant will attend the clinical investigation unit a 12 hour fast. A cannula will be placed in their forearm. Three fasting blood samples will be taken (-30, -15 and 0). A standard test meal of one Kellogg's breakfast bar and an Ensure Plus will be given. Blood will be taken at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180 amd 240 mins. This will be used to calculate Glucose profile, basal insulin response, dynamic phase insulin, static phase insulin sensitivity, DI=Dynamic phase insulin X Static phase insulin, GIP and GLP-1 response.

Free living glucose monitoring: Medtronic iPro Continuous Glucose Monitor will be used to assess 5-day continuous glucose monitoring. 5-day continuous glucose monitoring to assess "free living" glucose homeostasis. This interstitial fluid glucose data will be analysed for mean glucose and glycaemic variability measures including Mean Amplitude Glycaemic Excursions (MAGE), Continuous Overlapping Net Glycaemic Action (CONGA) and risk indices such as Low Blood Glucose Index (LBGI), High Blood Glucose Index (HBGI) and average daily risk ratio (ADRR). For the participant this will mean having a small plastic cannula place in the subcutaneous tissue in their abdomen. The participants will also be required to take 3 finger-prick glucose measurements on 4 successive days while wearing the CGM.

WHOLE BODY MRI SCANNING In investigation 3, whole body anatomical MR scanning will be performed to determine total and regional fat volumes, and magnetic resonance spectroscopy (MRS) performed to measure lipid content in the internal organs, such as liver (IHCL) and muscles (IMCL), such as soleus and tibialis.

Participants will attend the Robert Steiner MRI unit at Hammersmith Hospital after a 10h overnight fast. The study visit will last 1 hour. Participants are asked to refrain from strenuous exercise and drinking alcohol the day before each visit.

Firstly subjects will complete a metal check form. Next subjects will change into hospital clothes and be asked to lie on the trolley in the scanner. Subjects lie supine or prone in the scanner and are automatically moved through the scanner. While in the scanner participants will have access to a buzzer to sound an alarm, and will be able to hear and respond to instructions from the scanning console. Subjects will be in the MRI scanner for up to 1 hour. Scanning will be performed on either the Philips 3.0 Tesla or Philips 1.5 Tesla MR scanners in the Robert Steiner MRI Unit at the Hammersmith Hospital. None of the magnetic resonance imaging techniques to be used employs ionising radiation or intravenous contrast agents. Participants will also have their weight, height, waist and hip circumference recorded with a tape measure.

ELIGIBILITY:
Inclusion Criteria:

* Investigation 1 and 3: An oral glucose tolerance test diagnostic of impaired glucose tolerance as defined by the WHO as a fasting plasma glucose<7.0mmol/l and a 2-h plasma glucose ≥7.8 and <11.1mmol/l and/or impaired fasting glucose, defined by the American Diabetes Association as a fasting plasma glucose of >5.6 and <6.9mmol/L.
* Investigation 2: An oral glucose tolerance test diagnostic of impaired glucose tolerance as defined by the WHO as a fasting plasma glucose<7.0mmol/l and a 2-h plasma glucose ≥7.8 and <11.1mmol/l. For investigation 2, people with only IFG will be excluded.
* All investigations:
* Adults over 18 years of age
* Males and Females with a BMI between 25-35 kg/m2. The BMI range of between 25-35Kg/m2 has been chosen as this is the range that the majority of overweight people fall into (1). At this level of overweight and obesity there is an increase in the risk of type 2 diabetes. Above 40 kg/m2 there appears to be decreased success with lifestyle advice.
* The volunteers should have given full written consent.
* Have had a stable body weight for the last 6 months with no more than a 5% change in body weight over 6 months.

Exclusion Criteria:

* Adults less than 18 years of age.
* Volunteers with a major metabolic disease - including diabetes.
* A normal oral glucose tolerance test or that diagnostic of diabetes by the WHO criteria.
* Pregnant and lactating women.
* Males and Females with a BMI less than 25kg/m2 or greater than 35kg/m2
* Volunteers unable to give informed consent for themselves.
* Has lost or gained 5% of their normal body weight in the last 6 months.
* Has a known/diagnosed gastrointestinal problem such as inflammatory bowel disease, irritable bowel syndrome etc
* Failure of the medical examination for inclusion into the study
* Those with anaemia (Hb <10g/l)
* Drug or alcohol abuse in the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, PhD, Study Chair — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guess ND, Dornhorst A, Oliver N, Frost GS. A Randomised Crossover Trial: The Effect of Inulin on Glucose Homeostasis in Subtypes of Prediabetes. Ann Nutr Metab. 2016;68(1):26-34. doi: 10.1159/000441626. Epub 2015 Nov 17. PMID 26571012
- [Derived] Guess ND, Dornhorst A, Oliver N, Bell JD, Thomas EL, Frost GS. A randomized controlled trial: the effect of inulin on weight management and ectopic fat in subjects with prediabetes. Nutr Metab (Lond). 2015 Oct 24;12:36. doi: 10.1186/s12986-015-0033-2. eCollection 2015. PMID 26500686
- [Derived] Guess ND, Caengprasath N, Dornhorst A, Frost GS. Adherence to NICE guidelines on diabetes prevention in the UK: Effect on patient knowledge and perceived risk. Prim Care Diabetes. 2015 Dec;9(6):407-11. doi: 10.1016/j.pcd.2015.04.005. Epub 2015 May 13. PMID 25979539

RESULTS

PARTICIPANT FLOW:
Groups:
- Inulin: Inulin intervention
- Cellulose: Cellulose intervention
Period: Overall Study
Arm/Group | Inulin | Cellulose
Started | 22 | 22
Completed | 20 | 19
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Inulin: Participant received inulin
- Cellulose: Participants received cellulose
- Total: Total of all reporting groups
Arm/Group | Inulin | Cellulose | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12) | 59.7 (8.9) | 58.95 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 10 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 19 | 39
Weight [Mean (Standard Deviation); unit: kg] | 88.2 (14) | 83.4 (19.7) | 85.8 (16.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (4.1) | 30 (2.3) | 30.4 (3.2)
Haemoglobin A1c [Mean (Standard Deviation); unit: mmol/mol] | 5.9 (0.1) | 5.7 (0.1) | 5.8 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Glycaemic Control
Description: An oral glucose tolerance test (OGTT) using 75 g of glucose was performed to clarify glycaemic status.
Time Frame: 9 weeks
Measure: Mean (Standard Error); unit: mmol//l
Groups:
- Inulin: Received Inulin intervention
- Cellulose: Received Cellulose intervention
Arm/Group | Inulin | Cellulose
Number analyzed (Participants) | 20 | 19
mmol//l | -0.23 (0.17) | 0.44 (0.24)
Statistical Analysis 1: Comparison: Inulin vs Cellulose; Test type: Superiority; p = 0.005, ANCOVA — p-value was calculated, and is not attempting to indicate the threshold for statistical significance

2. Secondary Outcome: Food Intake in Gram at 9 Weeks
Description: Food intake following intervention over 9 weeks compared to baseline and between the two group
Time Frame: 9 weeks
Measure: Mean (Standard Error); unit: g
Arm/Group | Inulin | Cellulose
Number analyzed (Participants) | 20 | 19
g | -127 (45.4) | -0.47 (22.5)
Statistical Analysis 1: Comparison: Inulin vs Cellulose; Test type: Superiority; p = 0.027, ANCOVA

3. Other Pre Specified Outcome: Percentage Change in Body Weight
Description: Change in body weight over 9 week intervention
Time Frame: 9 weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Inulin | Cellulose
Number analyzed (Participants) | 20 | 20
percentage change | -5.3 (0.1) | -4.3 (0.4)
Statistical Analysis 1: Comparison: Inulin vs Cellulose; Test type: Superiority; p = 0.13, ANCOVA

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Inulin | Cellulose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes